CLINICAL TRIAL: NCT01309958
Title: Development of a Patient Based Provider Intervention for Early Caries
Brief Title: DPBRN Development of a Patient Based Provider Intervention for Early Caries Management
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Gregg H. Gilbert, DDS, MBA, FAAHD, Study Chair, University of Alabama at Birmingham, Dental Practice-Based Research Network
Other Study IDs: 018592; U01DE016747 (NIH)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Dental Caries
Keywords: Dental Caries; Intervention; Non-invasive treatment for early caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intervention: design instruments and test feasibility of an intervention aimed at increasing the proportion on non-invasive treatment for early caries

SUMMARY:
This study focused on improving the quality of dental care by fostering movement of the latest scientific advances into daily clinical practice.

DETAILED DESCRIPTION:
Phase 1 - development of two instruments (a patient brochure that described non-invasive caries treatment and a patient questionnaire of satisfaction with non-invasive caries treatment).

Phase 2 - field tested the patient brochure

Phase 3 - pilot tested the patient brochure, quantifying patient satisfaction with non-invasive caries treatments and a feasibility study that will inform the design of a clinical trial in dental practices envisioned for a later study.

ELIGIBILITY:
Inclusion Criteria:

* dentists enrolled in the Dental Practice-Based Research Network (DPBRN) who participated in DPBRN Assessment of Caries Diagnosis & Caries Treatment and DBPRN Reasons for placing the First Restoration on Permanent Tooth Surfaces

Exclusion Criteria:

* patients under 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ghg@uab.edu
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Gilbert, DDS, MBA, Principal Investigator — National Dental PBRN
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org
- See also: Dental Practice-Based Research Network — http://DPBRN.org